CLINICAL TRIAL: NCT02175979
Title: SANICS II Trial: A Multicenter Prospective Double-blind Randomized Controlled Trial Investigating the Effect of Stimulation of the Autonomic Nervous System in Colorectal Surgery by Perioperative Nutrition
Brief Title: SANICS II Trial: Stimulation of the Autonomic Nervous System in Colorectal Surgery by Perioperative Nutrition
Acronym: SANICSII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misha D.P. Luyer (Other)
Collaborators: Danone Global Research & Innovation Center (Industry); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Fonds NutsOhra (Other)
Responsible Party: Sponsor-Investigator, Misha D.P. Luyer, dr. M.D.P. Luyer, Catharina Ziekenhuis Eindhoven
Organization: Catharina Ziekenhuis Eindhoven (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL45640.060.13
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-08

CONDITIONS: Postoperative Ileus; Anastomotic Leak
Keywords: postoperative ileus; anastomotic leak; colorectal surgery; inflammation
MeSH Terms: conditions — Anastomotic Leak; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard (Placebo Comparator): standard of care
  Interventions: Dietary Supplement: standard
- enriched enteral nutrition (Experimental): enriched enteral tube feeding 1.5ml/ minute perioperative
  Interventions: Dietary Supplement: enriched enteral nutrition

INTERVENTIONS:
Dietary Supplement: enriched enteral nutrition — enriched enteral tube feeding perioperative
  Arms: enriched enteral nutrition
Dietary Supplement: standard — standard of care
  Arms: standard

SUMMARY:
The main objective is to investigate the effects of perioperative nutrition on postoperative ileus and anastomotic leakage in patients undergoing colorectal surgery.

Perioperative enteral nutrition is compared to the standard of care (fasting perioperatively).

DETAILED DESCRIPTION:
Postoperative ileus (POI) and anastomotic leakage (AL) are important clinical determinants of short-term morbidity and mortality following colorectal surgery. Importantly, AL is also a risk factor for local recurrence of colorectal cancer and has a significant impact on disease-free and overall survival. It is therefore believed that improving postoperative outcome following colorectal surgery will also improve long-term oncological outcomes regarding overall survival and tumour recurrence. POI is a common complication after colorectal surgery that causes discomfort for the patient but also leads to a prolonged hospital length of stay and increasing health care costs. For POI it is believed that formation of an inflammatory infiltrate in the muscular layers of the intestine following bowel manipulation during surgery leads to a decreased gastrointestinal motility. In recent years the investigators have demonstrated in experimental models that administration of enteral nutrition modulates the inflammatory response via the autonomic nervous system by release of cholecystokinin (CCK). Composition of the enteral nutrition and timing of administration are both essential for the magnitude of effect. For the most optimal effect, nutrition is given with a higher fraction of lipids and protein and is administered just before, during and directly after the inciting event. In this way, the inflammatory response is optimally dampened via release of CCK. In an experimental study has been shown that such a lipid-enriched enteral nutrition reduces systemic inflammation and postoperative ileus in a CCK-dependent manner when given just before and directly after bowel manipulation. Next, the investigators performed a study in healthy volunteers in which the effect of continuous low volume enteral nutrition was investigated on inflammatory parameters in a human endotoxemia model. In this study was shown that lipid enriched nutrition reduced the inflammatory response upon endotoxemia in man. Also in a clinical setting the investigators have shown that enteral nutrition reduces inflammation and postoperative ileus. In a randomized controlled trial the investigators have shown that enteral nutrition early after colorectal surgery reduced POI. Furthermore, in a model of sham-feeding using chewing gum was shown that inflammation and postoperative ileus were reduced following colorectal surgery. Interestingly, both clinical studies with sham feeding and early enteral nutrition revealed a yet unaccountable effect on anastomotic leakage. Evidence on the relation between POI and anastomotic leakage is scarce but has great impact. It seems that an early intervention with enteral nutrition shortly before, during and early after colorectal surgery may reduce inflammation and reduce important determinants in postoperative morbidity as POI and anastomotic leakage.

All patients will receive a self-migrating nasojejunal tube one day before surgery. The position of the nasojejunal tube is verified by means of an X-ray at the night before surgery. Preoperatively, patients receive standard of care with a fast for solid (oral) food of 6 hours and a (oral) fluid fast for 2 hours before administration. Three hours before surgery the pump is started to administer nutrition in standardized amounts. Enriched enteral nutrition (produced by Danone research) is administered via a programmed Flocare enteral feeding pump. The pump is connected to the opaque branched system that is connected both to the nasojejunal tube and to a sealed container. Patients are either allocated to the experimental group, in which the blinded branched system leads the enteral nutrition via the nasojejunal tube to the patient. Via this route, the patients in the experimental group will receive the enteral nutrition just before, during and directly after surgery. In patients allocated to the control group, the blinded branched system leads the enteral nutrition to the container. Consequently, when the feeding pump starts just before surgery, patients in the control group do not receive the nutrition. In both groups, the pump with enteral nutrition is stopped 6 hours after surgery and normal intake is resumed.

Based on previous results a power calculation is performed. For POI a sample size of at least 91 patients per group is needed based on a power of 0.8 and an alpha of 0.05. For AL a reduction of AL of at least 75% was observed in the previous clinical studies. Using a power of 0.8 and a drop-out percentage of 5% a total of 140 patients are needed per group. Since perioperative nutrition is a new concept, a safety analysis is performed after inclusion of 40 patients in which feasibility and safety of preoperative nutrition are assessed. The effect size is determined based on previous studies and is substantial. Considering the size of the effect, an interim-analysis will be performed after inclusion of 140 patients.

All analyses will be done according to the intention-to-treat approach in which all randomized patients are included, regardless of adherence to the study protocol. Occurrences of the primary and secondary endpoints are compared between the treatment groups. Results are presented as risk ratios with corresponding 95% confidence intervals. A two-tailed P < 0.05 is considered statistically significant. To compare the groups, the data will be tested for normal distribution and an unpaired T-test will be performed when appropriate, otherwise the Mann-Whitney U or Chi-square tests. SPSS (Statistical Package for the Social Sciences version 20) will be used to analyze the data.

The investigators respect the Dutch Scientific Code of conduct with regard to collection and storage of our data. The investigators hereby mind the criteria of retrievability, accessibility and interchangeability of the data. The investigators will obtain written informed consent from all patients, in which is stated that their records will be used and saved for research purposes for a minimum of 15 years. Anonymity and confidentiality of data will be guaranteed compliant with CBP (Commission Protection of Personal Data) guidelines. Thus, all variables will be registered anonymously, but via a secured code, personally identifiable information can be retrieved. The investigators verified completeness of patient Data Management Strategy via the Data Archiving and Networked Services checklist. Rough data will be stored in a digital archive, with appended description, to interpret the data.

ELIGIBILITY:
Inclusion Criteria:

* patients that undergo elective surgical resection of the colon or rectum with primary anastomosis.
* written informed consent
* age >18 years

Exclusion Criteria:

* use of medication that disrupts acetylcholine metabolism
* steroid use
* previous gastric or esophageal resection
* peritoneal metastases found during surgery
* ileostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-08; Primary Completion 2017-03-20 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Misha DP Luyer, MD PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (5):
- Denmark (2):
  - Regionshospitalet Randers, Randers
  - Regionshospitalet Viborg, Viborg
- Netherlands (3):
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Maxima Medical Center, Veldhoven, North Brabant
  - Elkerliek Ziekenhuis, Helmond

REFERENCES:
- [Background] Lubbers T, Luyer MD, de Haan JJ, Hadfoune M, Buurman WA, Greve JW. Lipid-rich enteral nutrition reduces postoperative ileus in rats via activation of cholecystokinin-receptors. Ann Surg. 2009 Mar;249(3):481-7. doi: 10.1097/SLA.0b013e318194d187. PMID 19247038
- [Background] Luyer MD, Greve JW, Hadfoune M, Jacobs JA, Dejong CH, Buurman WA. Nutritional stimulation of cholecystokinin receptors inhibits inflammation via the vagus nerve. J Exp Med. 2005 Oct 17;202(8):1023-9. doi: 10.1084/jem.20042397. Epub 2005 Oct 10. PMID 16216887
- [Background] Boelens PG, Heesakkers FF, Luyer MD, van Barneveld KW, de Hingh IH, Nieuwenhuijzen GA, Roos AN, Rutten HJ. Reduction of postoperative ileus by early enteral nutrition in patients undergoing major rectal surgery: prospective, randomized, controlled trial. Ann Surg. 2014 Apr;259(4):649-55. doi: 10.1097/SLA.0000000000000288. PMID 24169163
- [Background] Lubbers T, Kox M, de Haan JJ, Greve JW, Pompe JC, Ramakers BP, Pickkers P, Buurman WA. Continuous administration of enteral lipid- and protein-rich nutrition limits inflammation in a human endotoxemia model. Crit Care Med. 2013 May;41(5):1258-65. doi: 10.1097/CCM.0b013e31827c0a17. PMID 23388517
- [Background] Luyer MD, Habes Q, van Hak R, Buurman W. Nutritional stimulation of the autonomic nervous system. World J Gastroenterol. 2011 Sep 14;17(34):3859-63. doi: 10.3748/wjg.v17.i34.3859. PMID 22025873
- [Background] Luyer MD, Derikx JP, Beyaert R, Hadfoune M, van Kuppevelt TH, Dejong CH, Heineman E, Buurman WA, Greve JW. High-fat nutrition reduces hepatic damage following exposure to bacterial DNA and hemorrhagic shock. J Hepatol. 2009 Feb;50(2):342-50. doi: 10.1016/j.jhep.2008.08.025. Epub 2008 Nov 8. PMID 19070388
- [Background] Luyer MD, Buurman WA, Hadfoune M, Jacobs JA, Dejong CH, Greve JW. High-fat enteral nutrition reduces endotoxin, tumor necrosis factor-alpha and gut permeability in bile duct-ligated rats subjected to hemorrhagic shock. J Hepatol. 2004 Sep;41(3):377-83. doi: 10.1016/j.jhep.2004.04.026. PMID 15336439
- [Background] Luyer MD, Jacobs JA, Vreugdenhil AC, Hadfoune M, Dejong CH, Buurman WA, Greve JW. Enteral administration of high-fat nutrition before and directly after hemorrhagic shock reduces endotoxemia and bacterial translocation. Ann Surg. 2004 Feb;239(2):257-64. doi: 10.1097/01.sla.0000108695.60059.80. PMID 14745335
- [Derived] Peters EG, Smeets BJJ, Nors J, Back CM, Funder JA, Sommer T, Laurberg S, Love US, Leclercq WKG, Slooter GD, de Vries Reilingh TS, Wegdam JA, Nieuwenhuijzen GAP, Hiligsmann M, Buise MP, Buurman WA, de Jonge WJ, Rutten HJT, Luyer MDP. Perioperative lipid-enriched enteral nutrition versus standard care in patients undergoing elective colorectal surgery (SANICS II): a multicentre, double-blind, randomised controlled trial. Lancet Gastroenterol Hepatol. 2018 Apr;3(4):242-251. doi: 10.1016/S2468-1253(18)30031-1. Epub 2018 Feb 14. PMID 29426699
- [Derived] Peters EG, De Jonge WJ, Smeets BJ, Luyer MD. The contribution of mast cells to postoperative ileus in experimental and clinical studies. Neurogastroenterol Motil. 2015 Jun;27(6):743-9. doi: 10.1111/nmo.12579. PMID 26011782
- [Derived] Peters EG, Smeets BJ, Dekkers M, Buise MD, de Jonge WJ, Slooter GD, Reilingh TS, Wegdam JA, Nieuwenhuijzen GA, Rutten HJ, de Hingh IH, Hiligsmann M, Buurman WA, Luyer MD. The effects of stimulation of the autonomic nervous system via perioperative nutrition on postoperative ileus and anastomotic leakage following colorectal surgery (SANICS II trial): a study protocol for a double-blind randomized controlled trial. Trials. 2015 Jan 27;16:20. doi: 10.1186/s13063-014-0532-x. PMID 25623276

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard | Enriched Enteral Nutrition
Started | 140 | 140
Completed | 133 | 132
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Population: in both arms, 140 patients participated. in the standard arm 7 patients had to quit the study because exclusion criteria were met, in the enriched enteral nutrition 8 patients had to quit the study because exclusion criteria were met, which is stated in the results participant flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard | Enriched Enteral Nutrition | Total
Number analyzed (Participants) | 133 | 132 | 265
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [63 to 74] | 69 [62 to 75] | 68 [63 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 52 | 107
  Male | 78 | 80 | 158
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 101 | 103 | 204
  Denmark | 32 | 29 | 61
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 26 [24 to 29.3] | 25.8 [23.2 to 29] | 25.8 [23.7 to 29.1]
smoking currently [Count of Participants; unit: Participants] | 17 | 14 | 31
use of alcohol currently [Count of Participants; unit: Participants] | 92 | 100 | 192
use of neoadjuvant therapy for resection [Count of Participants; unit: Participants] | 20 | 27 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Developing Postoperative Ileus
Description: number of patients with absence of flatus or stool passage and inability to tolerate a regular oral diet between surgery and postoperative day 4
Time Frame: up to 3 weeks after surgery
Measure: Count of Participants; unit: Participants
Groups:
- Enriched Enteral Nutrition: enriched enteral tube feeding
Arm/Group | Standard | Enriched Enteral Nutrition
Number analyzed (Participants) | 133 | 132
Participants | 29 | 37

2. Secondary Outcome: Anastomotic Leakage
Description: number of patients developing anastomotic leakage
Time Frame: up to 6 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | Enriched Enteral Nutrition
Number analyzed (Participants) | 133 | 132
Participants | 11 | 12

3. Secondary Outcome: Aspiration Pneumonia
Description: number of patients developing aspiration pneumonia
Time Frame: up to 3 week after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | Enriched Enteral Nutrition
Number analyzed (Participants) | 133 | 132
Participants | 0 | 0

4. Secondary Outcome: Gastric Motility
Description: Percent change in Gastric Antral Area, assessed by Ultrasound of the Gastric Antrum Following a Standardized Meal
Time Frame: 3 days after surgery
Population: not every patients was fit to have the standard meal or ultrasound, therefore less antral measurements were executed.
Measure: Median (Inter-Quartile Range); unit: percentage of decrease in antral area
Arm/Group | Standard | Enriched Enteral Nutrition
Number analyzed (Participants) | 109 | 106
percentage of decrease in antral area | -32.7 [-45.9 to -9.2] | -31.4 [-46.6 to -9.8]

5. Secondary Outcome: Functional Recovery
Description: Length of functional recovery in days, Functional recovery was defined as postoperative patients not receiving intravenous fluid who have adequate pain control, restoration ofindependent mobility, sufficient caloric intake, and no signs of active infection
Time Frame: up to 6 weeks after surgery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard | Enriched Enteral Nutrition
Number analyzed (Participants) | 133 | 132
days | 5 [3 to 7] | 5 [3 to 9]

6. Secondary Outcome: C-reactive Protein (CRP)
Description: the inflammatory response measured systemically (in blood): C-reactive protein (CRP)
Time Frame: up to 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Standard | Enriched Enteral Nutrition
Number analyzed (Participants) | 113 | 114
mg/L | 150 [99 to 220] | 164 [108 to 227]

7. Secondary Outcome: Number of Patients Needing Additional Surgical, Radiological or Endoscopic Interventions
Description: number of patients needing additional surgical, radiological or endoscopic interventions: All surgical complications are classified using the Clavien-Dindo classification. patients with a Clavien Dindo grade IIIa, IIIb, IVa, IVb, V complication had a surgical, radiological or endoscopic intervention.
Time Frame: up to 6 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | Enriched Enteral Nutrition
Number analyzed (Participants) | 133 | 132
Participants | 21 | 15

8. Secondary Outcome: Number of Patients Needing ICU Admission
Description: number of patients needing ICU admission after surgery
Time Frame: up to 6 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | Enriched Enteral Nutrition
Number analyzed (Participants) | 133 | 132
Participants | 37 | 31

9. Secondary Outcome: Health-related Quality of Life
Description: Global Quality of life on a scale ranging from 0 to 100, with higher scores indicating higher level of functioning. The EORTC QLQ C-30 questionnaires are used
Time Frame: 6 months after surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard | Enriched Enteral Nutrition
Number analyzed (Participants) | 102 | 116
units on a scale | 83 [75 to 85] | 78 [67 to 83]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Standard | Enriched Enteral Nutrition
All-Cause Mortality (participants affected / at risk) | 7/133 | 4/132
Serious Adverse Events (participants affected / at risk) | 52/133 | 55/132
Other Adverse Events (participants affected / at risk) | 22/133 | 16/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard (N=133) | Enriched Enteral Nutrition (N=132)
anastomotic leakage (Gastrointestinal disorders) | 12 | 11
remaining serious adverse events (Surgical and medical procedures) | 40 | 44 — serious adverse events according to the official definition in the study protocol, not including the patients with anastomotic leakage
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard (N=133) | Enriched Enteral Nutrition (N=132)
clavien dindo grade 1 (Surgical and medical procedures) | 22 | 16 — clavien dindo grade 1: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT02175979/Prot_SAP_000.pdf